CLINICAL TRIAL: NCT02301494
Title: Feasibility Study to Determine Effectiveness of 3.75% Topical Imiquimod Cream and Topical Vanos (Fluocinonide) Cream 0.1% in the Treatment of Early Stage Cutaneous T-cell Lymphoma
Brief Title: Effectiveness of Imiquimod Topical Cream in Early Stage Cutaneous T-cell Lymphoma
Acronym: CTCL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled in the study.
Sponsor: Rochester General Hospital (Other)
Collaborators: Bausch Health Americas, Inc. (Industry); Rochester Skin Lymphoma Medical Group, PLLC (Other)
Responsible Party: Principal Investigator, Brian Poligone, MD, PhD, Scientist II, Rochester General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 48861
Record Dates: First submitted 2014-11-19; First posted 2014-11-26 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Mycosis Fungoides
Keywords: CTCL; Mycosis Fungoides; Cutaneous T-cell Lymphoma; MF; topical therapy; early stage
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous | interventions — Fluocinonide

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluocinonide (Vanos) cream 0.1% (Experimental): Fluocinonide (Vanos) cream 0.1% will be applied as currently approved by the FDA for treatment of corticosteroid responsive disorders of the skin. Treatment will continue for 4 months with a follow up at 6 and 12 months.
  Interventions: Drug: 0.1% Fluocinonide Cream
- 3.75% Imiquimod (Zyclara) Cream (Experimental): 3.75% Imiquimod (Zyclara) Cream will be used as currently labeled by the FDA for treatment of actinic keratoses. Treatment will continue for 4 months with follow up at 6 and 12 months.
  Interventions: Drug: 3.75% Imiquimod Cream

INTERVENTIONS:
Drug: 3.75% Imiquimod Cream — CTCL specific assessments to measure response in lesions will be done at each visit. Therapy initiates at day 1 followed by a visit at day 15. Visits will then be once a month for four months with a follow up at 6 and 12 months.
  Other Names: Zyclara 3.75%
  Arms: 3.75% Imiquimod (Zyclara) Cream
Drug: 0.1% Fluocinonide Cream — CTCL specific assessments to measure response in lesions will be done at each visit. Therapy initiates at day 1 followed by a visit at day 15. Visits will then be once a month for four months with a follow up at 6 and 12 months.
  Other Names: Vanos
  Arms: Fluocinonide (Vanos) cream 0.1%

SUMMARY:
This study is being conducted by Brian Poligone, MD PhD. The purpose of this study is to determine safety, effectiveness, and tolerability of two topical therapies, imiquimod and fluocinonide, for patients with early stage Cutaneous T-cell Lymphoma (CTCL).

DETAILED DESCRIPTION:
The purpose of the study is to compare the safety, effectiveness, and tolerability of two topical therapies, imiquimod and fluocinonide, for patients with early stage CTCL.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged ≥18 years.
2. Willing and able to give informed consent
3. Diagnosis of Mycosis Fungoides In cases with equivocal histological features, the diagnosis may be confirmed through the use of clonal T-cell gamma gene rearrangement, as detected by PCR amplification and primer sets specific for the T-cell receptor gamma chain genes.
4. Subjects must have at least one target lesion
5. Subjects will be able to comply with the study instructions, apply the study medication as directed and attend all visits.
6. Females of child-bearing potential must have a negative urine pregnancy test before randomization and must agree to use an adequate method of contraception (abstinence, condoms, hormonal therapy, barrier methods) during the study.
7. Patients must be otherwise healthy with an ECOG Performance status of 0 or 1.
8. The patient must not have had topical (2 weeks) or systemic therapy (4 weeks), radiotherapy (4 weeks) or phototherapy therapy (4 weeks) for Mycosis Fungoides within the stated number of weeks prior to start of treatment.
9. Eligible patients will be those who topical corticosteroid would be a preferred treatment and include patients newly diagnosed with stage IA, IB, or IIA disease, or those patients currently stable on therapy, in whom topical corticosteroids are being newly added to the regimen (i.e. recurrence or resistant lesions not currently treated with topical corticosteroids)

Exclusion Criteria:

To be eligible for inclusion in this study the subjects must not meet any of the following criteria:

1. Female who is pregnant, nursing an infant, or planning a pregnancy during the study period.
2. Have concomitant dermatologic or medical condition(s) which may interfere with the investigator's ability to evaluate the subject's response to the study drug.
3. Received any investigational drug or taking part in any clinical study within one month prior to this study.
4. Known reaction or allergy to test drug or excipient.
5. Presence of major medical illness or symptoms of a clinically significant illness that may influence the study.
6. Have any reason which, in the opinion of the investigator, interferes with the ability of the subject to participate in or complete the trial, or which places the subject at undue risk such as a history of drug, alcohol or other substance abuse or other factors limiting the ability to co-operate and to comply with this protocol.
7. Lesions on the genitals, axillae and face will not be selected for study treatment and evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Response Rate between baseline and week 16 | 16 weeks
  Treatment phase will last 4 months with follow up at 6 and 12 months after initiation of therapy

SECONDARY OUTCOMES:
Response Rate 24 and 52 weeks after baseline | Baseline to up to one year
  Patients will be treated for 4 months and response rate assessed at 6 and 24 months after initiation of therapy.
Safety and tolerabiliy of Imiquimod in patients with CTCL (adverse events) | From Randomization to up to 30 days after end of treatment
  We will record any adverse events that occur during the course of the study.
Learn about T cell dysregulation in the skin from patients with CTCL (Using left over tissue from biopsies) | Samples may be stored indefinitely from time of collection ( two weeks after initiation of therapy, and optional one done at week16)
  Using left over tissue from biopsies done at baseline, two weeks after initiation of therapy, and optional one done at week16. We are interested in making our tissue bank.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Poligone, M.D. Ph.D., Principal Investigator — Rochester General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956